CLINICAL TRIAL: NCT01671735
Title: VA Diabetes Prevention: Epidemiology of Pre-Diabetes and Implementation Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not considered a clinical trial because both treatment protocols have been approved as usual care
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRP 12-440
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes
Keywords: prevention; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VA DPP (Experimental): Pre-Diabetic Participants eligible for VA DPP receive a curriculum based life-style intervention program tailored off of the original DPP but in a group format
  Interventions: Other: Survey
- VA DPP-eligible MOVE! (No Intervention): Pre-Diabetic participants who screen and are eligible for VA DPP but bc of class being filled - have been assigned to MOVE!

INTERVENTIONS:
Other: Survey — A clinical demonstration project funded by NCP will involve screening Veterans and enrolling veterans with pre-diabetes into the VA DPP program. This research project will recruit VA DPP eligible participants enrolled in the VA DPP program and Veterans enrolled in MOVE! that are VA DPP eligible as a comparison group. The research is not truly an intervention but similar to a program evaluation.
  Arms: VA DPP

SUMMARY:
This study will collect baseline survey data from a NCP funded VA Diabetes Prevention Program (VA DPP) clinical demonstration program at three medical centers on VA DPP participants and VA DPP-eligible VA MOVE! participants to identify baseline participant demographic characteristics; attitudes and beliefs about diet, exercise and weight loss, and psychosocial constructs such as social support; and self-regulation skills that predict 6-month weight loss and program attendance. The data collected will contribute to our knowledge of pre-diabetic Veterans' attitudes and beliefs about diet, exercise and weight loss, to our understanding of how different programs may impact weight loss, and to evidence-based targeting in future clinical implementation projects. It will also provide baseline quality of life data for use in a future cost-effectiveness analysis.

DETAILED DESCRIPTION:
Background:

Type 2 diabetes is a preventable disease. Multiple large scale randomized controlled trials have shown that in people with impaired glucose tolerance, Type 2 diabetes can be prevented with prevention lifestyle interventions that emphasize diet, exercise and weight loss. The Diabetes Prevention Program (DPP) showed that lifestyle interventions can reduce the incidence of type 2 diabetes by 58% in this high risk group. Little is known about the incidence of pre-diabetes in the VA because routine screening for pre-diabetes is not an established practice in the VA. With a few exceptions, lifestyle modification interventions that target individuals with pre-diabetes and follow the Diabetes Prevention Program curriculum are not available to Veterans in the VA. In order to address this gap in evidence based clinical services, the National Center for Health Promotion and Disease Prevention (NCP) has funded a VA Diabetes Prevention Program Demonstration Project (VA DPP) at 3 VA Medical Centers (Baltimore, Minneapolis, and Greater Los Angeles). NCP has requested assistance to conduct a more extensive implementation focused evaluation of VA DPP.

Methods Baseline survey data will be collected from 720 Veterans eligible for the VA DPP (360 in the VA DPP group, 360 in VA MOVE!) from 3 Medical Centers across the country. All participants referred to the VA MOVE! program will be evaluated for VA DPP eligibility and scheduled for a VA MOVE! orientation meeting. At that face-to-face orientation meeting, VA DPP-eligible Veterans will be invited to complete the baseline survey after completing an informed consent process and signing a written informed consent document. Consented Veterans will be provided with a paper copy of the survey, a stamped return envelope addressed to the Ann Arbor VA coordinating center and an incentive gift card or voucher. Instructions on the survey will include a URL link to an online survey that can be used by Veterans who prefer to answer the survey online as opposed to taking the paper survey. The survey will include a unique participant code that will be used to match survey data with clinical and administrative data by participant. The participant code will also be used to access the online survey. There will be no other personal identifiers on the survey.

Objectives

1. To identify baseline participant demographic characteristics: attitudes and beliefs about diet, exercise and weight loss: psychosocial constructs such as social support; and self-regulation skills that predict 6-month weight loss and program attendance.
2. To collect baseline survey data on hypothesized modifiable mediators of program impact on weight loss including outcome expectations, self-regulation, skill mastery, willingness to self-monitor, self-efficacy for use in subsequent analyses after 6- and 12-month survey data and to collect quality of life data to be used in future cost-effectiveness studies.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese Veterans who qualify for VA MOVE! who also have pre-diabetes by the CDC
* NDPRP criteria (fasting glucose of 100 to 125 mg/dl or Hgb A1C of 5.7 to 6.4 )
* and who live within one hour of one of three VAMCs (Baltimore, Minneapolis and Greater Los Angeles) will be eligible for the VA DPP program
* Veterans who have been assigned to the VA DPP program or Veterans who have been screened for the VA DPP program are eligible but classes have been filled and have been assigned to VA MOVE! will be asked to consent to complete a survey questionnaire at the time of enrollment
* They will also be asked to consent for access to link their program data (such as weight, BMI, visit attendance) to their survey data

Exclusion Criteria:

* Patients with A1C of 6.5-6.9% although considered pre-diabetic by VA criteria, will be excluded, as they are considered diabetic based upon ADA and NDPRP criteria for the VA DPP clinical program
* Similarly, patients who are being treated with metformin will be excluded, to avoid confounding factors in the analysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
weight loss | one year

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Richardson, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States